CLINICAL TRIAL: NCT04850430
Title: Gastric Venous Reconstruction to Reduce Gastric Venous Congestion After Total Pancreatectomy
Brief Title: Gastric Venous Reconstruction After Total Pancreatectomy
Acronym: GENDER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Arianeb Mehrabi, MD, Professsor, Head of the Division of Liver Surgery and Visceral Transplantation, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-173/2021
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Pancreas Cancer; Pancreatectomy
Keywords: Pancreatectomy; Gastric venous outflow reconstruction; Gastric venous congestion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to study after intraoperative evaluation of gastric venous drainage after coronary vein resection during TP. During surgery, onsite evaluation by the surgeon, endoscopic examination, indocyanine green, gastric venous drainage flowmetry, and spectral analysis will be performed. After surgery, patients will receive standard post-TP care and treatment. During hospitalization, endoscopic examination with indocyanine green will be performed on the first, third, and seventh postoperative day to evaluate gastric ischemia. Ischemia markers will be evaluated daily after surgery. After discharge, patients will be followed up for 30 days, during which mortality and morbidities will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric venous congestion following total pancreatectomy (Experimental): The gastric venous outflow will be reconstructed after TP. The patients will be assessed concerning gastric venous congestion and gastric ischemia intraoperatively before and after venous outflow reconstruction through onsite evaluation by the surgeon, endoscopic examination, indocyanine green, gastric venous drainage flowmetry, and spectral imaging.
  Interventions: Procedure: Gastric venous reconstruction

INTERVENTIONS:
Procedure: Gastric venous reconstruction — Patients will be assigned to study after intraoperative evaluation of gastric venous drainage after coronary vein resection during TP, and the gastric venous outflow will be reconstructed after TP.

SUMMARY:
Total pancreatoduodenectomy (TP) is the standard surgical approach for treatment of extended pancreas tumors. If the gastric coronary vein has to be sacrificed for oncologic or for technical reasons in total pancreatectomy with splenectomy, gastric venous congestion (GVC) may result because all major venous draining routes are terminated. In the sequelae of GVC, gastric venous infarction ultimately leads to gastric perforation with abdominal sepsis. To avoid gastric venous infarction, partial or even total gastrectomy is usually performed in the event of GVC after TP. However, this significantly impacts the patient's quality of life.

Reconstruction of gastric venous outflow represents a technical approach to overcome GVC and to avoid gastric venous infarction making (partial) gastrectomy unnecessary. The current study aims to assess the role of gastric venous outflow reconstruction in GVC after TP to prevent (partial) gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provide written informed consent
* Elective total pancreatectomy for malignant or benign pancreatic lesions or chronic pancreatitis with splenectomy
* Intraoperative ligation of coronary vein

Exclusion Criteria:

* Gastric resection due to malignant infiltration
* Non-reconstructable gastric venous drainage
* Previous pancreas surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastric venous congestion | 30 days postoperative
  Gastric venous congestion after gastric venous reconstruction following total pancreatectomy
Incidence of gastric ischemia | 30 days postoperative
  Gastric ischemia after gastric venous reconstruction following total pancreatectomy
Postpancreatectomy gastrectomy rate | 30 days postoperative
  Rate of gastrectomy after gastric venous reconstruction following total pancreatectomy
Reoperation rate | 30 days postoperative
  Reoperation rate after gastric venous reconstruction following total pancreatectomy
Morbidity rate | 30 days postoperative
  Complications rate after gastric venous reconstruction following total pancreatectomy
Mortality rate | 30 days postoperative
  Mortality rate after gastric venous reconstruction following total pancreatectomy

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Surgery clinic, Heidelberg
  - Professor Dr. med. Arianeb Mehrabi, Heidelberg

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, the data generated by the current research that supports our future article, would be made available as soon as possible, wherever legally and ethically possible.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Mehrabi A, Loos M, Ramouz A, Dooghaie Moghadam A, Probst P, Nickel F, Schaible A, Mieth M, Hackert T, Buchler MW. Gastric venous reconstruction to reduce gastric venous congestion after total pancreatectomy: study protocol of a single-centre prospective non-randomised observational study (IDEAL Phase 2A) - GENDER study (Gastric vENous DrainagE Reconstruction). BMJ Open. 2021 Oct 21;11(10):e052745. doi: 10.1136/bmjopen-2021-052745. PMID 34675020